CLINICAL TRIAL: NCT03954132
Title: EVELUT®: Assessment of Dyspnea and Other Symptoms as Patient Reported Outcomes (PRO) in Patients With Chronic Obstructive Pulmonary Disease (COPD), Symptomatic on LABA/ICS Maintenance Therapy (Now) Treated With Spiolto® Respimat® (Tiotropium/Olodaterol) in Comparison to Open or Fixed Triple Combination Treatment in Routine Clinical Practice
Brief Title: Spiolto® Respimat® (Tiotropium/Olodaterol) Versus Triple Combination Therapy in Everyday Clinical Treatment Practice for Chronic Obstructive Pulmonary Disease (EVELUT®)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0087
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spiolto® Respimat®: Chronic Obstructive Pulmonary Disease (COPD) patients who were symptomatic (dyspneic) despite Long-acting beta2 adrenoceptor agonist/Inhalative Corticosteroids (LABA/ICS) maintenance treatment were switched to Spiolto® Respimat® inhaler by their attending physician in an real-world setting.
  Interventions: Drug: Spiolto® Respimat®
- Triple-Therapy (LAMA/LABA/ICS): Chronic Obstructive Pulmonary Disease (COPD) patients who were symptomatic (dyspneic) despite Long-acting beta2 adrenoceptor agonist/Inhalative Corticosteroids (LABA/ICS) maintenance treatment were switched to any triple therapy Long-acting muscarinic antagonist + Long-acting beta2 adrenoceptor agonist + Inhalative Corticosteroids (LAMA + LABA + ICS) by their attending physician in an real-world setting.
  Interventions: Drug: Triple-Therapy (LAMA/LABA/ICS)

INTERVENTIONS:
Drug: Spiolto® Respimat® — Chronic Obstructive Pulmonary Disease (COPD) patients who were symptomatic (dyspneic) despite Long-acting beta2 adrenoceptor agonist/Inhalative Corticosteroids (LABA/ICS) maintenance treatment were switched to Spiolto® Respimat® inhaler by their attending physician in an real-world setting.
  Groups: Spiolto® Respimat®
Drug: Triple-Therapy (LAMA/LABA/ICS) — Chronic Obstructive Pulmonary Disease (COPD) patients who were symptomatic (dyspneic) despite Long-acting beta2 adrenoceptor agonist/Inhalative Corticosteroids (LABA/ICS) maintenance treatment were switched to any triple therapy Long-acting muscarinic antagonist + Long-acting beta2 adrenoceptor agonist + Inhalative Corticosteroids (LAMA + LABA + ICS) by their attending physician in an real-world setting.
  Groups: Triple-Therapy (LAMA/LABA/ICS)

SUMMARY:
Open-label comparative multicentric cohort study in COPD patients with LABA/ICS, switched to either tiotropium/olodaterol and observed for 12 weeks approximately.

DETAILED DESCRIPTION:
COPD patients on LABA/ICS maintenance therapy with dyspnea (mMRC ≥ 1) and other symptoms (CATTM ≥ 10), who are switched to either Spiolto® Respimat® in the new reusable inhaler or any triple therapy (LAMA + LABA + ICS) as an open or fixed combination according to approved SmPCs at baseline at the discretion of their attending physician.

ELIGIBILITY:
Inclusion Criteria:

Patients can be included if all of the following criteria are met:

* Diagnosis of COPD
* Symptomatic (with regard to dyspnea (mMRC Dyspnea score ≥1) AND with regard to symptoms (CAT Score ≥10) at the same time)
* Patients on LABA/ICS maintenance therapy who are switched to Spiolto® Respimat® in the new reusable inhaler or a free/fixed triple combination of LABA + LAMA + ICS at Visit 1 at the discretion of the treating physician.
* Adults who are contractually capable and mentally able to understand and follow the instructions of the study personnel
* Male or female
* Patients aged ≥40 years of age
* Written informed consent prior to study participation
* The patient is willing and able to follow the procedures outlined in the protocol

Exclusion Criteria:

* Patients with contraindications acc. to SmPC
* Patients not on LABA/ICS maintenance treatment at visit 1, e.g., mono or dual bronchodilation only, ICS only, or a triple combination of LAMA + LABA + ICS (either as a fixed combination product or as separate components)
* Lack of informed consent
* Pregnant and/or lactating females
* Acute exacerbation of COPD (within 4 weeks prior to Visit 1)
* Frequently exacerbating patients, i. e. patients with ≥2 moderate exacerbations within the last 12 months or ≥1 exacerbation leading to hospitalization within the last 12 months
* Acute respiratory failure (pH <7,35 and/ or respiratory rate >30/min within 3 months prior to Visit 1)
* History or current diagnosis of asthma
* History or current diagnosis of asthma-COPD overlap
* History or current diagnosis of allergic rhinitis within the last 5 years
* History or current diagnosis of lung cancer within the last 5 years
* Participation in a parallel interventional clinical trial
* mild exacerbation: additional use of short-acting bronchodilators and treated by the patient without consulting a physician
* moderate exacerbation: treatment includes medical prescription of a systemic corticosteroid and/or antibiotic
* severe exacerbation: exacerbation leading to hospitalization

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study is based on newly collected data from approximately 900 COPD patients from 150 recruiting sites in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 469 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Marseille, 0049613277141881, Study Chair — andrea.marseille@boehringer-ingelheim.com
Locations (75):
- Germany (75):
  - Dr. Graubner, Bad Sachsa
  - Dr. Junggeburth, Bad Wörishofen
  - Dr. Heinz, Bergisch Gladbach
  - Praxis E. Hossbach, Berkatal
  - Praxis an der Oper, Berlin
  - Dr. Urban, Berlin
  - Praxis A.Sahan/S. Erbil-Sahan, Berlin
  - Dr. Kopf, Berlin
  - Dres. Pabst/Schlünz, Bonn
  - Dr. Schwittay, Böhlen B Leipzig
  - Dres. Bartels/Bartels, Breuberg
  - Dr. Grimm-Sachs, Bruchsal
  - Praxis B. Metzlaff, Büchen
  - Ambulantes Zentrum, Cottbus
  - Lungenzentrum Darmstadt, Darmstadt
  - Hausarzt Deggingen, Deggingen
  - Dres. Tietjens, Dortmund
  - Dr. Schwiese, Duisburg
  - Schwerpunktpraxis, Düsseldorf
  - Dr. Schmorell, Forchheim, Oberfr
  - Praxis A. Xanthopoulos, Fürstenwalde
  - Dr. Sommer, Garmisch-Partenkirchen
  - Dres. Ern/Trilling, Gelsenkirchen
  - Dr. Birkner, Gelsenkirchen
  - Praxis C. Staack/Z. Zadrozny, Gelsenkirchen
  - Das HausarztZentrum, Grafenrheinfeld
  - Dres. Coesfeld/Gams/Gams, Gütersloh
  - Pneumologicum Halle, Halle
  - MVZ Martha-Maria gGmbH, Halle
  - Dr. Knolinski, Hamburg
  - Dres. Kaase/Lepinat, Hamburg
  - Dr. Abenhardt, Heidelberg, Neckar
  - Dr. Koch, Heilbad Heiligenstadt
  - Dres Stolpe/ Roß, Ibbenbueren
  - Dres. Lehmann/Schulze und Partner, Jerichow
  - Dr. Beckmann, Kamen, Westf
  - Praxis G. Mohanty, Kamp-Lintfort
  - Dr. Auge, Koblenz Am Rhein
  - Dres. Lehmann/Schulze und Partner, Köthen
  - Dr. Pfitzer, Kronach, Oberfr
  - Dres. Alshut/Weberling, Lahnau
  - Dr. Einenkel, Leipzig
  - Dr. Geßner, Leipzig
  - Dr. Pitule, Ludwigshafen am Rhein
  - Dr. Hladik, Ludwigshafen am Rhein
  - Dr. Saur, Mannheim
  - Dres. Jerrentrup/Mronga, Marburg
  - Dr. Jansen, Menden (Sauerland)
  - Dr. Ingerl, Mosbach, Baden
  - Dr. Feimer, München
  - Thoraxzentrum Bez. Unterfranken, Münnerstadt
  - Praxis Th. Hagen, Neumarkt in der Oberpfalz
  - Praxis W. Wuttke, Nuremberg
  - Dr. Laser, Nürnberg, Mittelfr
  - MVZ OB-Sterkrade GmbH, Oberhausen, Rheinl
  - Dr. Müller, Potsdam
  - Dres. Hennig/Mikes, Radebeul
  - Dr. Dinh, Rathenow
  - Zentrum für Onkologie, Rostock
  - Lungenfachzentrum Rhein-Main, Rüsselsheim am Main
  - Lungenzentrum Schleswig, Schleswig
  - Dres. Korupp/Rose, Schweinfurt
  - Dr. Theuer, Seelow
  - Praxis S. Schmidt, Siegen
  - Dres. Knöbel und Partner, Straubing
  - Dr. Rother, Strausberg
  - Marienhospital Stuttgart, Stuttgart
  - Dr. Schmidt-Reinwald, Trier
  - Lungenzentrum Ulm, Ulm, Donau
  - Dres. Günther/Günther, Viernheim
  - Dres. Waltert/Esselmann, Warendorf
  - Dres. Herold/Kaa, Weißenburg I Bay
  - Dres. Fried/Rubin, Wiesbaden
  - Dr. Franz, Witten
  - Dr. Weber, Witten

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Buhl R, Dreher M, Mattiucci-Guehlke M, Emerson-Stadler R, Eckhardt S, Taube C, Vogelmeier CF. EVELUT(R): A Real-World, Observational Study Assessing Dyspnoea and Symptom Burden in COPD Patients Switched from LABA/ICS to LAMA/LABA or LAMA/LABA/ICS. Adv Ther. 2023 Jul;40(7):3263-3278. doi: 10.1007/s12325-023-02524-y. Epub 2023 May 31. PMID 37256536
- [Derived] Buhl R, Dreher M, Korn S, Taube C, Stock C, Zehendner CM, Kondla A, Vogelmeier CF. A Non-Interventional Study of Tiotropium/Olodaterol versus Any Triple Combination Therapy for Chronic Obstructive Pulmonary Disease: The EVELUT(R) Study Protocol. Int J Chron Obstruct Pulmon Dis. 2020 Oct 22;15:2601-2608. doi: 10.2147/COPD.S262746. eCollection 2020. PMID 33122898
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label comparative multicentric cohort non interventional study based on newly collected data. Chronic Obstructive Pulmonary Disease (COPD) patients receiving a Long-acting beta2 adrenoceptor agonist/Inhalative Corticosteroids treatment until visit 1 were switched at the discretion of the attending physician to either tiotropium/olodaterol in the new reusable Respimat® inhaler or any triple therapy according to clinical routine. Observational period was approximately 12 weeks.
Pre-assignment Details: All patients were screened for eligibility prior to participation in the trial. 6 patients were not recruited and treated. 24 patients in the treated set had at least one violations of the in- and/or exclusion criteria and were not included in the per protocol set (and the derived matched set).
Period: Overall Study
Arm/Group | Spiolto® Respimat® | Triple-Therapy (LAMA/LABA/ICS)
Started (Patients with Visit 1 and treated (=Treated Set)) | 329 | 134
Per Protocol Set | 309 | 129
Treated Subjects With Protocol Violations (Treated patients with protocol violations, patients were excluded from the per protocol set.) | 19 | 5
Treated Subjects Excluded From Per Protocol Set (Patient excluded from per protocol set due to open query related to in-/exclusion criteria.) | 1 | 0
Completed (Patients with Visit 2) | 303 | 129
Not Completed | 26 | 5
Not completed — Adverse Event | 2 | 0
Not completed — Patient's wish | 5 | 0
Not completed — Lost to Follow-up | 10 | 0
Not completed — Screening failure | 0 | 1
Not completed — No registration after Visit 1 | 5 | 2
Not completed — Other reason than listed | 2 | 2
Not completed — Patient could not make visit due to vertebral fracture | 1 | 0
Not completed — False inclusion, violation of exclusion criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All patients with informed consent who have received at least one dose of Spiolto® Respimat® or triple combination (free or fixed LAMA + LABA+ ICS).
Groups:
- Total: Total of all reporting groups
Arm/Group | Spiolto® Respimat® | Triple-Therapy (LAMA/LABA/ICS) | Total
Number analyzed (Participants) | 329 | 134 | 463
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (10.7) | 69.2 (8.9) | 67.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 56 | 215
  Male | 170 | 78 | 248
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
modified Medical Research Council (mMRC) score [Mean (Standard Deviation); unit: Score on a scale] — The modified Medical Research Council (mMRC) scale is a 5-point (0-4) scale based on the severity of dyspnoea, where a 0 is the best possible score with no disability and 4 is the worst possible score representing the most severity. The mMRC will be used to assess the breathlessness state of the patient with just one question: "When do you experience dyspnoea?", covering five everyday activities, potentially leading to dyspnoea and giving an according rate of 0 to 4 points. Population: Matched set (MS): All patients with informed consent who met all inclusion criteria as well as no exclusion criteria and have received at least one dose of Spiolto® Respimat® or triple combination (free or fixed LAMA + LABA+ ICS), excluding all patients who could not be matched in the propensity score matching, patients with missing data were not replaced or imputed.
  Score on a scale
    number analyzed (Participants) | 121 | 121 | 242
    (all) | 2.07 (0.80) | 2.07 (0.81) | 2.07 (0.80)
CATᵀᴹ (COPD assessment test) score [Mean (Standard Deviation); unit: Score on a scale] — The Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CATᵀᴹ). The CATᵀᴹ consists of eight items, each formatted as a semantic six-point differential scale. These eight items cover cough, phlegm, chest tightness, breathlessness when going up hills/stairs, activity limitations at home, confidence leaving home, sleep and energy. Each item is scored from 0 to 5. Total CAT score is calculated as the sum over the 8 items, resulting in a total score ranging from 0 to 40, corresponding to the best and worst health status in patients with COPD, respectively. Population: Matched set (MS): All patients with informed consent who met all inclusion criteria as well as no exclusion criteria and have received at least one dose of Spiolto® Respimat® or triple combination (free or fixed LAMA + LABA+ ICS), excluding all patients who could not be matched in the propensity score matching, patients with missing data were not replaced or imputed.
  Score on a scale
    number analyzed (Participants) | 121 | 121 | 242
    (all) | 21.72 (6.29) | 21.79 (6.72) | 21.76 (6.49)

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Medical Research Council (mMRC) Score Between Baseline and After End of Observation
Description: Change in mMRC (modified Medical Research Council) score between baseline and after end of observation (ca. 12 weeks of treatment, Visit 2). The modified Medical Research Council (mMRC) scale is a 5-point (0-4) scale based on the severity of dyspnoea, where a 0 is the best possible score with no disability and 4 is the worst possible score representing the most severity. The mMRC will be used to assess the breathlessness state of the patient with just one question: "When do you experience dyspnoea?", covering five everyday activities, potentially leading to dyspnoea and giving an according rate of 0 to 4 points. The Minimum Clinically Important Difference (MCID) is a change of 1.0 point. Change calculated as Visit 1 - Visit 2.
Time Frame: Baseline at Visit 1 (day 0) and Visit 2 (planned at 12 week, up to a maximum of 42 weeks).
Population: Matched set (MS): All patients with informed consent who met all inclusion criteria as well as no exclusion criteria and have received at least one dose of Spiolto® Respimat® or triple combination (free or fixed LAMA + LABA+ ICS), excluding all patients who could not be matched in the propensity score matching, patients with missing data for this outcome measure were not replaced or imputed.
Measure: Mean (95% Confidence Interval); unit: Change in score on a scale
Groups:
- Spiolto® Respimat®, Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto): Chronic Obstructive Pulmonary Disease (COPD) patients who were symptomatic (dyspneic) despite Long-acting beta2 adrenoceptor agonist/Inhalative Corticosteroids (LABA/ICS) maintenance treatment were switched to Spiolto® Respimat® inhaler by their attending physician in an real-world setting. Patients were propensity score matched to the Triple-Therapy arm, propensity score was calculated based on a logistic regression model taking the choice of treatment as dependent variable and baseline characteristics as independent variables into account.
- Triple-Therapy (LAMA/LABA/ICS), Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto): Chronic Obstructive Pulmonary Disease (COPD) patients who were symptomatic (dyspneic) despite Long-acting beta2 adrenoceptor agonist/Inhalative Corticosteroids (LABA/ICS) maintenance treatment were switched to any triple therapy Long-acting muscarinic antagonist + Long-acting beta2 adrenoceptor agonist + Inhalative Corticosteroids (LAMA + LABA + ICS) by their attending physician in an real-world setting. Patients were propensity score matched to the Spiolto® Respimat® arm, propensity score was calculated based on a logistic regression model taking the choice of treatment as dependent variable and baseline characteristics as independent variables into account.
Arm/Group | Spiolto® Respimat®, Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto) | Triple-Therapy (LAMA/LABA/ICS), Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto)
Number analyzed (Participants) | 111 | 118
Change in score on a scale | 0.23 [0.11 to 0.36] | 0.25 [0.13 to 0.38]

2. Primary Outcome: Change in CATᵀᴹ (COPD Assessment Test) Score Between Baseline and After End of Observation (ca. 12 Weeks of Treatment)
Description: The Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CATᵀᴹ) was developed as a simple instrument to assess health status in patients with COPD. The CATᵀᴹ consists of eight items, each formatted as a semantic six-point differential scale, making the tool easy to administer and easy for patients to complete. These eight items cover cough, phlegm, chest tightness, breathlessness when going up hills/stairs, activity limitations at home, confidence leaving home, sleep and energy. Each item is scored from 0 to 5. Total CAT score is calculated as the sum over the 8 items, resulting in a total score ranging from 0 to 40, corresponding to the best and worst health status in patients with COPD, respectively. The Minimum Clinically Important Difference (MCID) is a change of 2.0 points. Change is calculated as Visit 1 - Visit 2.
Time Frame: Baseline at Visit 1 (day 0) and Visit 2 (planned at 12 week, up to a maximum of 42 weeks).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Change in score on a scale
Arm/Group | Spiolto® Respimat®, Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto) | Triple-Therapy (LAMA/LABA/ICS), Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto)
Number analyzed (Participants) | 111 | 118
Change in score on a scale | 3.45 [2.45 to 4.45] | 2.51 [1.62 to 3.40]

3. Secondary Outcome: Patients' General Condition According to the Physician's Global Evaluation (PGE) Score at Baseline
Description: The treating physician used the Physician's Global Evaluation (PGE) to evaluate the general condition of the patient on an 8-point ordinal scale from 1-2 (poor), 3-4 (satisfactory), 5-6 (good) to 7-8 (excellent).
Time Frame: Baseline at Visit 1 (day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®, Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto) | Triple-Therapy (LAMA/LABA/ICS), Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto)
Number analyzed (Participants) | 121 | 121
Participants
  PGE score 1 | 0 | 0
  PGE score 2 | 3 | 4
  PGE score 3 | 17 | 26
  PGE score 4 | 48 | 49
  PGE score 5 | 27 | 26
  PGE score 6 | 20 | 12
  PGE score 7 | 4 | 3
  PGE score 8 | 1 | 0
  Missing | 1 | 1

4. Secondary Outcome: Patients' General Condition According to the Physician's Global Evaluation (PGE) Score at the End of the Observation Period
Description: The treating physician will use the Physician's Global Evaluation (PGE) to evaluate the general condition of the patient on an 8-point ordinal scale from 1 (very poor) to 8 (excellent).
Time Frame: Visit 2 (planned at 12 week, up to a maximum of 42 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®, Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto) | Triple-Therapy (LAMA/LABA/ICS), Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto)
Number analyzed (Participants) | 112 | 119
Participants
  PGE score 1 | 0 | 1
  PGE score 2 | 3 | 3
  PGE score 3 | 9 | 18
  PGE score 4 | 27 | 31
  PGE score 5 | 26 | 25
  PGE score 6 | 34 | 28
  PGE score 7 | 12 | 9
  PGE score 8 | 1 | 2
  Missing | 0 | 2

5. Secondary Outcome: Patient Satisfaction With Inhaler and Therapy at End of Observation Period
Description: Patient satisfaction with inhaler and therapy at end of observation period according to a seven-point ordinal scale (ranging from very dissatisfied to very satisfied).
Time Frame: Visit 2 (planned at 12 week, up to a maximum of 42 weeks).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®, Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto) | Triple-Therapy (LAMA/LABA/ICS), Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto)
Number analyzed (Participants) | 112 | 55
Participants
  Patient overall satisfaction with treatment: Very satisfied | 31 | 17
  Patient overall satisfaction with treatment: Satisfied | 58 | 21
  Patient overall satisfaction with treatment: Rather satisfied | 7 | 7
  Patient overall satisfaction with treatment: Neither satisfied nor dissatisfied | 7 | 4
  Patient overall satisfaction with treatment: Rather dissatisfied | 4 | 2
  Patient overall satisfaction with treatment: Dissatisfied | 1 | 0
  Patient overall satisfaction with treatment: Very dissatisfied | 3 | 1
  Patient overall satisfaction with treatment: Missing | 1 | 3
  Patient satisfaction with handling of the inhalation device: Very satisfied | 27 | 17
  Patient satisfaction with handling of the inhalation device: Satisfied | 66 | 26
  Patient satisfaction with handling of the inhalation device: Rather satisfied | 11 | 5
  Patient satisfaction with handling of the inhalation device: Neither satisfied nor dissatisfied | 5 | 3
  Patient satisfaction with handling of the inhalation device: Rather dissatisfied | 2 | 0
  Patient satisfaction with handling of the inhalation device: Dissatisfied | 0 | 0
  Patient satisfaction with handling of the inhalation device: Very dissatisfied | 0 | 0
  Patient satisfaction with handling of the inhalation device: Missing | 1 | 4
  Patient satisfaction with inhaling from the device: Very satisfied | 31 | 20
  Patient satisfaction with inhaling from the device: Satisfied | 63 | 22
  Patient satisfaction with inhaling from the device: Rather satisfied | 8 | 6
  Patient satisfaction with inhaling from the device: Neither satisfied nor dissatisfied | 7 | 3
  Patient satisfaction with inhaling from the device: Rather dissatisfied | 2 | 0
  Patient satisfaction with inhaling from the device: Dissatisfied | 0 | 0
  Patient satisfaction with inhaling from the device: Very dissatisfied | 0 | 0
  Patient satisfaction with inhaling from the device: Missing | 1 | 4
  Patient satisfaction with the device in general: Very satisfied | 30 | 16
  Patient satisfaction with the device in general: Satisfied | 65 | 26
  Patient satisfaction with the device in general: Rather satisfied | 9 | 4
  Patient satisfaction with the device in general: Neither satisfied nor dissatisfied | 4 | 4
  Patient satisfaction with the device in general: Rather dissatisfied | 2 | 1
  Patient satisfaction with the device in general: Dissatisfied | 0 | 0
  Patient satisfaction with the device in general: Very dissatisfied | 1 | 0
  Patient satisfaction with the device in general: Missing | 1 | 4

6. Secondary Outcome: Number of Responders With Δ mMRC≥ 1
Description: Number of responders with a change in modified Medical Research Council (mMRC) greater than or equal to 1 between visit 1 and 2. The mMRC was used to assess the severity of the breathlessness. the mMRC consists of five statements describing the patients grade of breathlessness ranging from 0 (best outcome) to 4 (worst outcome).
Time Frame: Baseline at Visit 1 (day 0) and Visit 2 (planned at 12 week, up to a maximum of 42 weeks).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®, Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto) | Triple-Therapy (LAMA/LABA/ICS), Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto)
Number analyzed (Participants) | 112 | 119
Participants
  Δ mMRC<1 | 83 | 92
  Δ mMRC≥1 | 28 | 26
  Not available | 1 | 1

7. Secondary Outcome: Number of Responders With Δ CAT≥ 2
Description: Number of responders with a change in the Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) greater than or equal to 2 between visit 1 and 2.
Time Frame: Baseline at Visit 1 (day 0) and Visit 2 (planned at 12 week, up to a maximum of 42 weeks).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®, Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto) | Triple-Therapy (LAMA/LABA/ICS), Propensity Score Matched 1(Triple-Therapy) to 1(Spiolto)
Number analyzed (Participants) | 112 | 119
Participants
  Δ CAT<2 | 35 | 51
  Δ CAT≥2 | 76 | 67
  Not available | 1 | 1

ADVERSE EVENTS:
Time Frame: The study design is of non-interventional nature and the study is conducted within the conditions of the approved marketing authorization. Sufficient data from controlled interventional trials are available to support the evidence on the safety and efficacy of the studied BI drug. Collected were: - all adverse drug reaction (ADRs) (serious and non-serious), - all adverse events with fatal outcome
Description: From the beginning of treatment till the end of the study, up to 42 weeks.
Arm/Group | Spiolto® Respimat® | Triple-Therapy (LAMA/LABA/ICS)
All-Cause Mortality (participants affected / at risk) | 0/329 | 0/134
Serious Adverse Events (participants affected / at risk) | 1/329 | 0/134
Other Adverse Events (participants affected / at risk) | 0/329 | 0/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiolto® Respimat® (N=329) | Triple-Therapy (LAMA/LABA/ICS) (N=134)
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
There are some limitations due to the observational, non-randomized study concept. Imbalances between treatment groups could be due to the observational, non-randomized study design reflecting real-world data.

Less patients than originally planned have been included (900 patients planned vs. 469 patients actual). Patient inclusion was impaired by the Corona pandemic from early spring 2020 on.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT03954132/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT03954132/SAP_001.pdf